CLINICAL TRIAL: NCT04749563
Title: A Phase I Randomized Placebo Controlled MAD Study to Evaluate Safety and Tolerability of IGC-AD1 in Subjects With Dementia Due to Alzheimer's Disease
Brief Title: Study of IGC-AD1 in Subjects With Dementia Due to Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IGC Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: P1 IGC-AD1 BPSD
Record Dates: First submitted 2020-12-29; First posted 2021-02-11 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Dementia of Alzheimer Type

STUDY DESIGN:
Intervention Model Description: 3 dose escalation cohorts in same 12 subjects (5:1 randomization (active:placebo)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study subjects will be blinded to the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): IGC AD1
  Interventions: Drug: IGC AD1
- Placebo (Placebo Comparator): IGC AD1 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IGC AD1 — IGC AD1 oral Solution
  Arms: Active
Drug: Placebo — Placebo of IGC AD1 oral Solution
  Arms: Placebo

SUMMARY:
A single center, randomized, placebo controlled multiple ascending dose study of IGC AD1 to evaluate safety and tolerability in subjects with dementia due to Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This is a phase I Multiple Ascending Dose (MAD) study to evaluate safety and tolerability of IGC-AD1 in subjects with AD. Twelve subjects will be enrolled. Three different ascending doses of the study product will be given: low, medium and high doses. Each dose will be given for 2 weeks, followed by a washout period of 4 days. Given the vulnerability of the population, a safety cohort of 3 patients (2 active, 1 placebo) will start every dose one day ahead of the rest of the patients and will be followed for 24 hours for the development of Adverse Events (AEs). Objective criteria will be set after the safety cohort is evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and/or study partner (relative) must provide a signed and dated Informed Consent form prior to any study procedures which will be discussed with the Study Coordinator.
2. Provision of a letter from the Neurologist/Psychiatrist/Internal Medicine Physician certifying the diagnosis of Alzheimer's Dementia and patient's ability to consent. If patient is unable to consent, only the legal guardian/tutor of the patient could consent in his/her behalf. The guardian/tutor will be required to present the pertinent legal documentation.
3. Must have a study partner who is able and willing to comply with all required study procedures.
4. Patient should meet NIA-AA criteria for Alzheimer's disease, any stage.
5. At least 3 months evolution of behavioral symptoms at screening visit.
6. Negative drug screen, except for benzodiazepines if patient has been using them in stable doses for at least 3 months before screening.
7. All medications used for behavioral symptoms should be in stable doses for at least 3 months before screening.
8. All medications used for other conditions besides behavioral symptoms should be at stable doses for at least 30 days before screening.
9. Women must be postmenopausal (defined as cessation of menses for at least 1 year) or surgically sterile (hysterectomy, oophorectomy or bilateral tubal ligation) at the time of screening.

Exclusion Criteria:

1. Prior adverse reaction to cannabinoids.
2. Prior contraindication or allergy to any component of study product (IGC-AD1): melatonin, honey, curcumin, ethyl alcohol, vitamin-E TPGS, ascorbic acid, water, tween-80, and rutin.
3. History of stroke, multiple sclerosis (MS), or epilepsy. History of gastrointestinal dysfunction not related to Alzheimer's disease (e.g., inflammatory bowel disease or gastrointestinal cancer)
4. Any clinically relevant neurological disorder capable of producing a dementia syndrome including Parkinson's disease, stroke, vascular dementia, dementia with Lewy bodies, frontotemporal dementia, and others.
5. Other possible causes of dementia as: infections of the CNS (e.g. HIV, syphilis) or Creutzfeldt Jakob disease, subdural hematoma, communicating hydrocephalus, brain tumors, drug intoxication, alcohol intoxication, thyroid disease, parathyroid disease, and vitamin B12 or other deficiencies
6. Use of contraindicated medication (see section 6).
7. History of myocardial infarction, severe congestive heart failure, unstable angina, significant valvular disease, or cardiomyopathy within 1 year of screening.
8. History of cardiac arrhythmias, second or third-degree AV block.
9. History of seizures, schizophrenia, or bipolar disorder.
10. Other condition or clinically important abnormality on vital signs, physical examination, neurologic examination, laboratory results or electrocardiogram (ECG) examination that could compromise the study efficacy interpretation or safety of the subject.
11. Have participated in an investigational drug or device study within 30 days prior to study start.
12. TCA or opioid use within 30 days before the enrollment.
13. History of alcohol and drug abuse within 2 years of screening.
14. Elevated liver enzymes (AST or ALT ≥3 times upper limit of normal, Total bilirubin≥1.5 times ULN or ALP≥1.5 times ULN).
15. Urine drug screen positive for drug use, except for benzodiazepines if patient was using them previously and their dose had remained stable for at least 3 months before screening

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events in IGC-AD1 as compared to placebo [Safety and Tolerability] | 3 weeks
  Evaluate safety and tolerability of IGC AD1 10 participants will be administered the investigational drug and two will be administered placebo. Incidence of treatment emergent adverse events will be assessed to determine safety and tolerability of IGC-AD1.

SECONDARY OUTCOMES:
Measurement of efficacy using Neuropsychiatric Inventory (NPI) scale | 3 weeks
  Secondary Outcome: Comparison of the measurement of Neuropsychiatric Inventory (NPI) scale changes from baseline using the Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: IGC Pharma INC, Study Director — IGC Pharma INC
Locations (1):
- Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No